CLINICAL TRIAL: NCT01997684
Title: Colonic Stenting With Elective Surgery Versus Emergency Surgery in the Management of Acute Malignant Colonic Obstruction: a Multicentre, Prospective, Open Label, Cohort Study
Brief Title: Colonic Stenting With Elective Surgery Versus Emergency Surgery in the Management of Acute Malignant Colonic Obstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISR-ENDO-2013-001
Record Dates: First submitted 2013-11-18; First posted 2013-11-28 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Acute Malignant Colonic Obstruction; Colorectal Cancer; Colonic Obstruction
Keywords: Colorectal Cancer; Colonic Obstruction
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Elective Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colonic Stenting with Elective Surgery (Experimental): In the experimental group, the patients will undergo colonic stenting within 24 h of inclusion. For this study, the WallFlex ™ Colonic Stent (Boston Scientific, Natick, MA) will be employed.
  Candidates for elective surgery, after clinical success of colonic stenting, will be preferably operated on 5-14 days after inclusion, and no later than 4 weeks. Type and extent of the elective surgery will be selected by the surgeon.
  In this group, unplanned emergency surgery will be indicated in case of technical failure of colonic stenting, iatrogenic morbidity, or clinical failure.
  In case of a primary colostomy, restoration of bowel continuity was attempted within 3-6 months.
  Interventions: Procedure: Colonic Stenting with Elective Surgery
- Emergency Surgery (Active Comparator): In the comparator group, patients will be undergo emergency surgery. Surgical options including but not limited to: loop colostomy, Hartmann's procedure, and (sub) total colectomy with ileostomy or ileorectal anastomosis.
  In case of a primary colostomy, restoration of bowel continuity was attempted within 3-6 months.
  Interventions: Procedure: Emergency Surgery

INTERVENTIONS:
Procedure: Colonic Stenting with Elective Surgery — After preparation of the distal colon with an enema, the colonoscope will be introduced up to the site of the obstruction. The colonic stent will be placed along a guide wire through the lesion under radiologic or endoscopic guidance. A colonic stent will be chosen which was at least 3 cm longer than the lesion (1.5 cm at either end). When the colonic stent did not cover the entire length of the lesion, a second overlapping stent will be placed.
  If the colonic stenting failed (technical failure) or symptoms of colonic obstruction did not resolve within 3 days (clinical failure), patients were indicated for emergency surgery.
  Candidates for elective surgery were preferably operated on 5-14 days after colonic stenting, and no later than 4 weeks.
  Type and extent of the surgery were selected by the surgeon, including but not limited to: loop colostomy, Hartmann's procedure, and (sub) total colectomy with ileostomy or ileorectal anastomosis.
  Other Names: Colonic stenting as a bridge to elective surgery; Colonic stenting and elective surgery; Colonic stenting and deferred surgery; Preoperative colonic stenting
  Arms: Colonic Stenting with Elective Surgery
Procedure: Emergency Surgery — Type and extent of the surgery were selected by the surgeon, including but not limited to: loop colostomy, Hartmann's procedure, and (sub) total colectomy with ileostomy or ileorectal anastomosis.
  Arms: Emergency Surgery

SUMMARY:
The use of colonic stenting with elective surgery has been suggested as an alternative management for acute malignant colonic obstruction, as emergency surgery has a high risk of morbidity and mortality.

However, the available body of literature addressing their benefit in this setting is contradictory.

The purpose of this study is to determine the efficacy and safety of colonic stenting with elective surgery versus emergency surgery in the management of acute malignant colonic obstruction.

DETAILED DESCRIPTION:
Colorectal cancer is one commonly diagnosed malignancy worldwide, with an estimated 10 million new cases and 6 million deaths . Around 8%-29% of patients with colorectal cancer present with acute colonic obstruction, and 70% of all malignant obstruction occurs in the left-sided colon. It has been reported that about 15%-20 % of patients with colorectal cancer present with acute obstructive symptoms at the time of diagnosis.

Conventionally, these patients are treated with emergency surgery to restore luminal continuity, which includes a variety of strategies such as the so-called two-stage surgery involving primary resection with colostomy (i.e., Hartmann's procedure) or proximal colostomy followed by resection, and one-stage surgery involving primary resection with anastomosis. Whatever the strategy chosen, the emergency surgery has an associated high risk of morbidity and mortality, and about two-thirds of such patients end up with a permanent stoma, which caused lower health-related quality of life and costs associated with stoma care.

Since 1991, the colonic stenting has been applied as palliative treatment for patients with unresectable colorectal cancer. In 1993, Tejero et al. reported using colonic stenting as a bridge to definitive surgery. Recently, Zhang et al. conducted a meta-analysis of 8 studies (6 retrospective and 2 randomized trials) and indicated that stent placement before elective surgery, also known as a bridge to surgery, lead to a reduction in need of intensive care (risk ratio [RR], 0.42; 95% confidence interval, 0.19-0.93), stoma creation (RR, 0.70; 0.50-0.99), and overall complications (RR, 0.42; 0.24-0.71) compared with the emergency surgery cohort, meanwhile, colonic stenting with elective surgery achieved higher primary anastomosis rate (RR, 1.62; 1.21-2.16), and did not adversely affect the mortality and long-term survival. The most common complications of colonic stenting were re-obstruction (12%), migration (11%), and perforation (4.5%).

However, the available body of literature addressing the benefit of colonic stenting with elective surgery is contradictory, and limited by the lack of the prospective randomised controlled trials. Therefore, we plan to conduct this multicenter, prospective, open label,cohort study, to determine the efficacy and safety of colonic stenting with elective surgery versus emergency surgery in the management of acute malignant colonic obstruction.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age.
* Symptoms of colonic obstruction, existing less than one week.
* Malignant obstruction in the colon.
* Signed informed consent.

Exclusion Criteria:

* Severe cardio-pulmonary disease or other serious disease leading to unacceptable surgical risk.
* Patients with signs of peritonitis, perforation, sepsis, or other serious complications demanding emergency surgery.
* Patients with distal rectal cancer less than 8 cm from the anal verge.
* Patients with suspected or proven metastatic adenocarcinoma.
* Patients with unresectable colorectal cancer, or planning for palliative treatment.
* Previous colonic surgery.
* Pregnancy or lactation women, or ready to pregnant women.
* Not capable of filling out questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Rates of primary colorectal anastomosis | From date of randomization until the first follow-up ended, assessed up to 30 days
  The primary colorectal anastomosis was defined as: the patients received one-stage surgery and colorectal anastomosis by whatever elective or emergency surgery.

SECONDARY OUTCOMES:
Stoma rates | From date of randomization until the follow-up ended, assessed up to 2 years
  The stoma constructed for any reason, whether temporary or definitive.
Mortality | From date of randomization until the date of death from any cause, assessed up to 2 years
  Death from any cause.
Procedure related complication | From date of randomization until the first follow-up ended, assessed up to 30 days
  Including but not limited to: anastomotic leakage, wound infection, intra-abdominal sepsis, re-obstruction, stent migration, perforation, bleeding, etc.
Re-operation rates | From date of randomization until the follow-up ended, assessed up to 2 years
  Re-operation is defined as repeat surgery or endoscopic treatment for whatever reason within 2 years.
R0 resection | From date of randomization until the first follow-up ended, assessed up to 30 days
  R0 resection is defined as negative resection margins and no residual tumor.
Quality of life | From date of randomization until the follow-up ended, assessed up to 2 years
  Quality of life assessments will be done with the European Organisation for Research and Treatment of Cancer (EORTC) core questionnaire,EORTC QLQ-C30, and the questionnaire module for colorectal cancer, EORTC QLQ-CR29.
Hospital stay and cost | From date of the admission to discharge, assessed up to 30 days
Recurrence of colorectal cancer | From date of randomization until the follow-up ended, assessed up to 2 years

OTHER OUTCOMES:
Technical success | From date of randomization until the first follow-up ended, assessed up to 30 days
  Technically success is defined as successful endoscopic placement of the stent in the correct position.
Clinical success | From date of randomization until the first follow-up ended, assessed up to 30 days
  Clinical success is defined as the resolution of obstructive symptoms and the production of flatus or stool within 3 days after colonic stenting.

CONTACTS AND LOCATIONS:
Overall Officials: Side Liu, M.D., Study Chair — Department of Gastroenterology, Nanfang Hospital, Southern Medical University
Locations (9):
- China (9):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Guangdong Province Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Xiangya hospital central-south university, Changsha, Hunan
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Renji Hospital, Medical College of Shanghai Jiao Tong University, Shanghai, Shanghai Municipality

REFERENCES:
- [Background] van Hooft JE, Bemelman WA, Oldenburg B, Marinelli AW, Lutke Holzik MF, Grubben MJ, Sprangers MA, Dijkgraaf MG, Fockens P; collaborative Dutch Stent-In study group. Colonic stenting versus emergency surgery for acute left-sided malignant colonic obstruction: a multicentre randomised trial. Lancet Oncol. 2011 Apr;12(4):344-52. doi: 10.1016/S1470-2045(11)70035-3. PMID 21398178
- [Background] Pirlet IA, Slim K, Kwiatkowski F, Michot F, Millat BL. Emergency preoperative stenting versus surgery for acute left-sided malignant colonic obstruction: a multicenter randomized controlled trial. Surg Endosc. 2011 Jun;25(6):1814-21. doi: 10.1007/s00464-010-1471-6. Epub 2010 Dec 18. PMID 21170659
- [Background] Ghazal AH, El-Shazly WG, Bessa SS, El-Riwini MT, Hussein AM. Colonic endolumenal stenting devices and elective surgery versus emergency subtotal/total colectomy in the management of malignant obstructed left colon carcinoma. J Gastrointest Surg. 2013 Jun;17(6):1123-9. doi: 10.1007/s11605-013-2152-2. Epub 2013 Jan 29. PMID 23358847
- [Background] Cheung HY, Chung CC, Tsang WW, Wong JC, Yau KK, Li MK. Endolaparoscopic approach vs conventional open surgery in the treatment of obstructing left-sided colon cancer: a randomized controlled trial. Arch Surg. 2009 Dec;144(12):1127-32. doi: 10.1001/archsurg.2009.216. PMID 20026830
- [Background] Alcantara M, Serra-Aracil X, Falco J, Mora L, Bombardo J, Navarro S. Prospective, controlled, randomized study of intraoperative colonic lavage versus stent placement in obstructive left-sided colonic cancer. World J Surg. 2011 Aug;35(8):1904-10. doi: 10.1007/s00268-011-1139-y. PMID 21559998
- See also: Homepage of Nanfang Hospital, Southern Medical University — http://www.nfyy.com/
- See also: Homepage of Department of Gastroenterology, Nanfang Hospital, Southern Medical University — http://www.xhbnet.com/